CLINICAL TRIAL: NCT04492007
Title: Feasibility Testing of Patient Reported Outcomes - Informed Symptom Management System (PRISMS)
Acronym: PRISMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LCCC1929; R01NR016990 (NIH)
Record Dates: First submitted 2020-06-24; First posted 2020-07-30 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; Bladder Cancer; Ovarian Cancer; Cervical Cancer; Uterine Cancer
Keywords: ostomy (colostomy, urostomy, and ileostomy); symptom; self-management; caregiving; family research; telehealth; self-efficacy; quality of life; post-treatment care transition
MeSH Terms: conditions — Colorectal Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISMS (Experimental): In addition to usual care, participants assigned to this arm will have access to our Patient-Reported Outcomes-Informed Symptom Management System (PRISMS) program.
  Interventions: Behavioral: Patient-Reported Outcomes-Informed Symptom Management System (PRISMS)
- Usual Care (No Intervention): Participants assigned to this arm will receive the standard of care that is provided to all patients.

INTERVENTIONS:
Behavioral: Patient-Reported Outcomes-Informed Symptom Management System (PRISMS) — Participants will receive personalized self-care information and guidance based on their symptoms and signs of complications (e.g., skin infection, fatigue) from the web-based telehealth PRISMS program. They will also have access through this website a peer support online forum that is moderated by a research nurse as well as professional support through videoconferencing/telephone from the research nurse and also their healthcare providers at the hospital(s) if they experience moderate to severe symptoms and/or abnormal sign (e.g., body temperature is greater than 98.6 C
  Arms: PRISMS

SUMMARY:
This is a proof-of-concept pilot randomized clinical trial to test the feasibility of the innovative Patient-Reported Outcomes-Informed Symptom Management System (PRISMS) to enhance personalized supportive care for cancer patients and caregivers during post-treatment care transition.

DETAILED DESCRIPTION:
In this proof-of-concept study, our multidisciplinary team will conduct a pilot randomized clinical trial to test the feasibility of the innovative Patient-Reported Outcomes-Informed Symptom Management System (PRISMS) to enhance personalized supportive care for cancer patients and caregivers during post-treatment care transition. We will randomly assign 21 cancer patients with newly created ostomies for cancer treatment with curative intent and their primary caregivers to the PRISMS or usual care groups (21 patient-caregiver dyads, a total of 42 individuals). PRISMS is defined as a personalized psychoeducational website including monitoring and personal feedback. We will conduct pre- and post-assessments of QOL and PRO (symptoms) at baseline upon enrollment and 2 months later.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

* have been surgically treated for colorectal, bladder, ovarian, cervical, or uterine cancer with curative intent;
* be within one month of hospital discharge of a newly created ostomy with curative intent;
* be able to read and speak English;
* be 18 years or older;
* have a caregiver who is willing to participate in the study;

Caregivers must:

* be 18 years or older;
* be able to read and speak English;
* be identified as the primary caregiver by the patient;
* have not themselves been diagnosed with cancer or received cancer treatment during the study (to ensure that patients and caregivers focus their efforts on care of the patient).

Exclusion Criteria:

Patients and their caregivers will be excluded if they:

* are unable to read, speak, or understand English;
* have more than one type of ostomy;
* have other cancer diagnosis (excluding non-melanomatous skin cancer); or
* have cognitive impairment (assessed by the Short Portable Mental Status Questionnaire).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Song, RN, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study with very small sample size and specific inclusion criteria. Sharing data with others may increase the risk to patient confidentiality.

REFERENCES:
- [Derived] Xu S, Tan X, Ma C, McElyea RS, Shieh K, Stover AM, Smith A, Stitzenberg K, Basch E, Song L. An eHealth symptom and complication management program for cancer patients with newly created ostomies and their caregivers (Alliance): a pilot feasibility randomized trial. BMC Cancer. 2023 Jun 10;23(1):532. doi: 10.1186/s12885-023-10919-x. PMID 37301841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study between 11/02/2020 - 8/10/2021 at one cancer center in North Carolina.
Pre-assignment Details: In total 46 participants, 23 patients, and 23 patients' caregivers were started to the study. Patients and their caregivers were graded as dyed; 16 dyed in the PRISM arm and 7 dyed in the control arm were enrolled in the study.
Groups:
- Caregiver-Usual Care: The primary caregiver of the participants assigned to this arm will receive the standard of care that is provided to all patients.
- PRISMS: Participants will receive personalized self-care information and guidance based on their symptoms and signs of complications from the web-based telehealth PRISMS program. They will also have access through this website a peer support online forum that is moderated by a research nurse as well as professional support through video conferencing/telephone from the research nurse and also their healthcare providers at the hospital(s).
- Caregiver-PRISMS: The primary caregiver of the participants assigned to receive eceive personalized self-care information and guidance based on their symptoms and signs of complications from the web-based telehealth PRISMS program. They will also have access through this website a peer support online forum that is moderated by a research nurse as well as professional support through video conferencing/telephone from the research nurse and also their healthcare providers at the hospital(s).
Period: Overall Study
Arm/Group | Usual Care | Caregiver-Usual Care | PRISMS | Caregiver-PRISMS
Started | 7 | 7 | 16 | 16
Completed | 5 | 5 | 12 | 12
Not Completed | 2 | 2 | 4 | 4
Not completed — Lost to Follow-up | 1 | 1 | 2 | 2
Not completed — Protocol Violation | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Subjects started to study interventions.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Caregiver-Usual Care | PRISMS | Caregiver-PRISMS | Total
Number analyzed (Participants) | 7 | 7 | 16 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.71 (25.81) | 38.00 (27.47) | 56.81 (13.73) | 48.06 (16.30) | 51.04 (19.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 4 | 11 | 24
  Male | 5 | 0 | 12 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 16 | 16 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 2 | 8
  White | 5 | 5 | 12 | 13 | 35
  More than one race | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 16 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Number
Description: The enrollment rate is defined as the number of potentially eligible couples (dyads) who have consented to participate in the study. 1 Dyad = 1 participant + their caregiver. Potentially eligible dyads (subjects and their caregivers) were approached and informed about the study. then the number of dyads who consented and completed.
Time Frame: Baseline
Population: Potentially eligible dyads (subjects and their caregivers) were approached and informed about the study. A total of 29 dyads were approached and were eligible and 25 dyads were consented.
Measure: Number; unit: Number of dyad participants
Groups:
- Potentially Eligible Dyads Recruited Into The Study: The number of Dyads successfully consented and completed the baseline survey among all people approached for the study.
Arm/Group | Potentially Eligible Dyads Recruited Into The Study
Number analyzed (Participants) | 29
Number of dyad participants | 25

2. Primary Outcome: Number of Potentially Eligible Dyads Participants Actually Enrolled in the Study
Description: Potentially Eligible Dyads Participants Actually Enrolled in the Study will be evaluated by the number of dyads who successfully consented and completed the baseline survey among all people approached for the study. 1 Dyad = 1 participant + their caregiver.
Time Frame: Baseline, after consent
Population: 25 dyads were consented.
Measure: Number; unit: Number of dyad participants
Groups:
- Percentage of Potentially Eligible Participants Recruited Into The Study: Percentage of patients participants and their caregivers successfully consented and completed the baseline survey among all people approached for the study.
Arm/Group | Percentage of Potentially Eligible Participants Recruited Into The Study
Number analyzed (Participants) | 25
Number of dyad participants | 23

3. Primary Outcome: Number of Dyads Remained in the Study and Completed the Post-Intervention Follow-Up Survey.
Description: The number of dyad Participants Enrolled who Remained in the Study and Completed the Post-Intervention Follow-Up Survey was assessed by the number of enrolled dyad participants who completed the 2-month follow-up survey at the end of the study period.
Time Frame: Up to 3 months (2-month follow up survey)
Population: The number of dyads who started to study completed baseline and post-intervention survey. Twenty-five dyads consented, and 23 of them completed the baseline survey.
Measure: Number; unit: Number of dyad participants
Groups:
- Potentially Eligible Participants Recruited Into The Study: Percentage of patients participants and their caregivers successfully consented and completed the baseline survey among all people approached for the study.
Arm/Group | Potentially Eligible Participants Recruited Into The Study
Number analyzed (Participants) | 23
Number of dyad participants | 17

4. Primary Outcome: Usability of Reported Outcomes - Patient Reported Outcomes - Informed Symptom Management System (PRISMS)
Description: Usability of Reported Outcomes - Patient Reported Outcomes - Informed Symptom Management System (PRISMS) evaluates three aspects: General, content, and navigation, contains 19 items on a 5-point Likert scale, where 1 is "strongly disagree" and 5 is "strongly agree". The score for each aspect was calculated as the sum of the scores from all items in this aspect. The scores ranged between 5 and 25 for General and Content, and the Navigation score ranged between 9 and 45. The higher score of the specific aspect that patients and their caregivers reported indicates the better usability of the aspect. This survey was offered separately at the follow-up visit to patients and their caregivers. Participants who completed at least 80.00% of the questions were included in the analysis. Usual Care and Informed Symptom Management System (PRISMS) group scores were compared.
Time Frame: Up to 2 months (Follow up survey)
Population: Thirty -four participants (17 patients and 17 caregivers) who completed the survey questionnaires were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Usual Care Patient: Patient participants assigned to this arm will receive the standard of care that is provided to all patients.
- Usual Care- Caregivers: Caregivers of patient participants assigned to this arm will receive the standard of care that is provided to all patients.
- PRISMS Patients: Patient participants will receive personalized self-care information and guidance based on their symptoms and signs of complications from the web-based telehealth PRISMS program. They will also have access through this website to a peer support online forum that is moderated by a research nurse as well as professional support through video conferencing/telephone from the research nurse and also their healthcare providers at the hospital(s).
- PRISMS- Caregivers: Caregivers of patient participants will receive personalized self-care information and guidance based on their symptoms and signs of complications from the web-based telehealth PRISMS program. They will also have access through this website to a peer support online forum that is moderated by a research nurse as well as professional support through video conferencing/telephone from the research nurse and their healthcare providers at the hospital(s).
Arm/Group | Usual Care Patient | Usual Care- Caregivers | PRISMS Patients | PRISMS- Caregivers
Number analyzed (Participants) | 5 | 5 | 12 | 12
score on a scale
  general aspect | 17.00 (3.65) | 17.50 (2.07) | 20 (3.66) | 20.36 (3.20)
  content aspect | 19.75 (4.99) | 18.50 (3.11) | 20.71 (3.41) | 21.36 (3.83)
  navigation aspect | 35.69 (7.46) | 37.45 (7.24) | 38.16 (6.37) | 30.75 (1.89)

5. Primary Outcome: Satisfaction With the PRISMS Program
Description: The satisfaction survey evaluates satisfaction with various aspects, contains 9 items on a 5-point Likert scale of 1 to 5, and higher scores reflect better satisfaction. Questions: Q1. The amount of time to review the program every time. Q2. Ease of navigating. Q3. Information I received. Q4. Quality of the information I received. Q5. The program has increased my knowledge about managing my symptoms and complications. Q6. The program has improved how I manage my symptoms and complications. Q7. The program has improved how I communicate with my family about sensitive topics related to my cancer care. Q8. The time and effort took me to complete. Q9. My knowledge about how my cancer has affected my partner and our relationship was improved. This survey was offered at the follow-up visit to patients and their caregivers separately. More than 80.00% of the questions answered were included in the analysis. The mean score for each question for Usual Care and PRISMS were compared.
Time Frame: 2-month followup survey
Population: Thirty -four participants (17 patients and 17 caregivers) who completed the survey questionnaires were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PRISMS -Caregivers: Caregivers of patient participants will receive personalized self-care information and guidance based on their symptoms and signs of complications from the web-based telehealth PRISMS program. They will also have access through this website to a peer support online forum that is moderated by a research nurse as well as professional support through video conferencing/telephone from the research nurse and their healthcare providers at the hospital(s).
Arm/Group | Usual Care | Usual Care- Caregivers | PRISMS | PRISMS -Caregivers
Number analyzed (Participants) | 5 | 5 | 12 | 12
score on a scale
  Q1 | 3.20 (1.10) | 3.20 (1.48) | 4.08 (0.79) | 3.83 (0.72)
  Q2 | 3.60 (1.34) | 4.20 (0.84) | 4.08 (1.00) | 4 (0.95)
  Q3 | 3.40 (1.14) | 4.00 (1.00) | 4.00 (0.95) | 3.92 (0.90)
  Q4 | 3.60 (0.89) | 4.20 (1.1) | 4.08 (1.00) | 4 (0.85)
  Q5 | 3.80 (1.10) | 3.60 (1.14) | 4.08 (1.00) | 4.17 (0.72)
  Q6 | 3.60 (0.89) | 3.40 (1.52) | 3.75 (1.22) | 4.17 (0.72)
  Q7 | 3.40 (0.89) | 3.60 (1.14) | 3.17 (1.40) | 4.00 (0.95)
  Q8 | 3.20 (1.48) | 2.40 (1.14) | 3.83 (1.19) | 3.64 (1.12)
  Q9 | 3.80 (0.84) | 3.60 (1.67) | 3.64 (1.29) | 3.92 (0.79)

6. Secondary Outcome: Difference of Quality of Life Change Over Time as Assessed by The Functional Assessment of Cancer Therapy - General (FACT-G).
Description: Quality of Life Change Over Time as Assessed by The Functional Assessment of Cancer Therapy - General (FACT-G) at baseline and follow-up visit to patients and their caregivers separately. Change from baseline is the post-baseline value minus the Baseline value. FACT-G is a 27-item survey that assesses physical, social/family, emotional, and functional well-being on a 5-point Likert scale, with 0 indicating "not at all" and 4 indicating "very much" in response to item questions. The total FACT-G score is calculated as the sum of four sub-scores including physical, social/family, emotional, and functional well-being. Total scores range between 0-108. Higher scores indicated better well-being. It has also demonstrated sensitivity to change over time Mean FACT-G difference between baseline and 2 months were presented.
Time Frame: baseline , 2 months
Population: Thirty -four participants (17 patients and 17 caregivers) who completed the survey questionnaires were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Usual Care- Caregivers | PRISMS | PRISMS- Caregivers
Number analyzed (Participants) | 5 | 5 | 12 | 12
score on a scale | 18.43 (13.59) | 13.57 (33.64) | 7.41 (8.98) | 9.53 (13.86)

7. Secondary Outcome: Difference of Anxiety Change Over Time as Assessed by PROMIS-Emotional Distress-Anxiety Short Form 7a
Description: Difference of Anxiety Change Over Time as Assessed by PROMIS-Emotional Distress-Anxiety Short Form 7a used to examine the change in anxiety among patients and their caregivers separately, from Baseline to follow up (2 months).
  For all PROMS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The anxiety sub-scale of the PROMIS item bank measures the extent to which participants experience anxiety symptoms over the past 7 days using a 5-point Likert scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with the total scores range from 36.3 to 82.7 with higher scores reflect higher anxiety.
Time Frame: Baseline and 2 months
Population: Thirty -four participants (17 patients and 17 caregivers) who completed the survey questionnaires were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PRISMS - Caregivers: Caregivers of patient participants will receive personalized self-care information and guidance based on their symptoms and signs of complications from the web-based telehealth PRISMS program. They will also have access through this website to a peer support online forum that is moderated by a research nurse as well as professional support through video conferencing/telephone from the research nurse and their healthcare providers at the hospital(s).
Arm/Group | Usual Care | Usual Care- Caregivers | PRISMS | PRISMS - Caregivers
Number analyzed (Participants) | 5 | 5 | 12 | 12
score on a scale | 6.56 (1.55) | 10.02 (8.48) | 13.42 (3.59) | 13.22 (3.62)

8. Secondary Outcome: Difference of Depression Change Over Time as Assessed by PROMIS-Emotional Distress-Depression Short From 8b
Description: Change of Depression Change Over Time as Assessed by PROMIS-Emotional Distress-Depression Short From 8b will be assessed by PROMIS-Emotional Distress-Depression Short From 8b. It is used to measure the change in depression scores among patients and their partners from Baseline (T1) to T2 (2 months post-T1). Required by the PROMIS scoring instrument, for all PROMS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The depression sub-scale of the PROMIS item bank measures the extent to which participants experience depressive symptoms in the past 7 days using a 5-point Likert scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with the total scores range from 24.7 to 63.5 with higher scores indicate greater depressive symptoms.
Time Frame: Baseline, 2 months
Population: Participants who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | PRISMS
Number analyzed (Participants) | 5 | 12
score on a scale
  Patients | 14.77 (8.83) | 8.55 (4.76)
  Patients' caregiver | 20.94 (5.60) | 11.08 (1.63)

9. Secondary Outcome: Difference Pain Score Over Time as Assessed by PROMIS Pain Interference - Short Form 6b
Description: Change Pain Score Over Time as Assessed by PROMIS Pain Interference - Short Form 6b will be assessed by PROMIS Pain Interference - Short Form 6b. It is used to measure the change in Pain. It was offered to patients and their caregivers separately. Required by the PROMIS scoring instrument, for all PROMS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The pain measures the extent to which patients experience problems with pain over the past 7 days using a 5-point Likert scale. Higher scores reflect greater Pain Interference. The score value ranges between 41-78.3.
Time Frame: Baseline, 2 months
Population: Thirty -four participants (17 patients and 17 caregivers) who completed the survey questionnaires were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Usual Care- Caregivers | PRISMS | PRISMS -Caregivers
Number analyzed (Participants) | 5 | 5 | 12 | 12
score on a scale | 7.28 (13.00) | 24.85 (5.28) | 13.02 (2.39) | 7.72 (15.60)

10. Secondary Outcome: Difference of Fatigue Change Over Time as Assessed by PROMIS Fatigue -Short Form 7a
Description: PROMIS Fatigue -Short Form 7a is used to measure the change in Fatigue among patients and their caregivers separately, from Baseline (T1) to T2 (2 months post-T1). Required by the PROMIS scoring instrument, for all PROMS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The fatigue scale measures the extent to which patients and their partners experience problems with fatigue over the past 7 days using a 5-point Likert scale. Higher scores reflect greater fatigue. Score value ranges between 29.4 - 83.2.
Time Frame: Baseline, 2 months
Population: Thirty -four participants (17 patients and 17 caregivers) who completed the survey questionnaires were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Usual Care- Caregivers | PRISMS | PRISMS - Caregivers
Number analyzed (Participants) | 5 | 5 | 12 | 12
score on a scale | 8.73 (29.94) | 46.19 (6.18) | 10.86 (7.48) | 16.28 (5.76)

11. Secondary Outcome: Change in Sleep Among Caregivers.
Description: Change in Sleep among caregivers. was assessed by the 22-item version of the Zarit Burden Interview is a caregiver self-reported instrument. It is used to assess caregiving burden change among caregivers from Baseline (T1) to T2 (2 months post-T1). Each item on the interview is a statement that the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Higher scores reflect more severe burden, 0-21: no to mild burden; 21-40: mild to moderate burden; 41-60: moderate to severe burden; ≥ 61: severe burden. The score value ranges between 0-88.
Time Frame: Baseline, 2 months
Population: Patients' caregivers participants responded to the survey questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | PRISMS
Number analyzed (Participants) | 5 | 12
score on a scale | 16.49 (29.84) | 0.40 (11.15)

ADVERSE EVENTS:
Time Frame: Not available, Adverse Events were not collected.
Description: The protocol does not require Adverse Event Collections and/or All-Cause Mortality data. Deaths and adverse events were not assessed.Since this study is a minimum risk educational intervention study. No Adverse Event happened during the study.
Arm/Group | Usual Care | Caregiver-Usual Care | PRISMS | Caregiver-PRISMS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators' joint publication is required.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT04492007/Prot_SAP_000.pdf